CLINICAL TRIAL: NCT03371290
Title: Acute Effect of Mirror Therapy on Motor Control, Manual Dexterity and Spasticity of Paretic Upper Extremity After Chronic Stroke
Brief Title: Acute Effect of Mirror Therapy on Rehabilitation of Paretic Upper Extremity After Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Caren Luciane Bernardi, Doctor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CEP UFCSPA 90050-170
Record Dates: First submitted 2017-11-27; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy Intervention (Experimental)
  Interventions: Other: Mirror Therapy
- Control Intervention (Active Comparator)
  Interventions: Other: Control Intervention

INTERVENTIONS:
Other: Mirror Therapy — The healthy UE will be positioned in front of the mirror and the paretic UE behind it, enabling the patient to observe the movements of the healthy limb through the mirror, interpreting that image as the affected limb. The MT protocol will be composed of active bimanual exercises of range of motion and functional exercises. Three sets of 15 repetitions will be performed for each exercise with a 20 seconds interval between each series, for 30 minutes. The exercises: 1) Elbow flexion/extension; 2) Wrist flexion/extension in neutral position; 3) Fingers flexion/extension in neutral position; 4) Forearm pronation/supination; 5) Roll the ball with hands; 6) Squeezing the sponge; 7) Drag a towel in anteroposterior direction; 8) Opponency of fingers; 9) Climb the mirror with the fingers (similar to walking the spider).
  Arms: Mirror Therapy Intervention
Other: Control Intervention — In the control intervention, patients will be performed the same bimanual activities proposed by the MT protocol, but without the reflector side of the mirror. The mirror will be placed in the same position as the MT intervention. However, the subject will have access to the non-reflective side of the mirror, directly visualizing the movement of his healthy arm.
  Both interventions will be performed a single session of MT or control composed of 30 minutes of exercises. The participants who will be first assigned to the MT intervention, after 4-weeks washout period, will be performed the same procedures, but in the control intervention. Likewise, patients who will be first allocated to control intervention, after 4-weeks of washout, will be performed the same procedures, however in MT intervention.
  Arms: Control Intervention

SUMMARY:
Objective: To investigate the acute effect of mirror therapy (MT) on motor control, manual dexterity and spasticity of the paretic upper extremity (UE) of individuals with chronic hemiparesis after stroke, during reaching task.

Design: Randomized cross-over single-blinded trial. Subjects: Thirty-three patients post chronic stroke were recruited of the study.

Intervention: Patients who first participated in the MT intervention performed a single session of MT, whereas in the control intervention a single session composed of the same exercises was performed, but without the mirror. After a month washout, the patients switched groups.

Main measure: The primary outcome measure was motor control. The secondary outcome measure was manual dexterity and UE spasticity.

The data will be expressed as mean and 95% confidence interval (continuous variable) and absolute frequency (categorical variables). To compare the outcomes of the different experimental sessions and at the different moments (pre and post session), the Generalized Estimating Equations with post hoc LSD (Least Significant Difference) methods will be used. For all analysis the significance level was set at α = 0.05 and statistical software SPSS (Statistical Package for Social Sciences for Mac, version 22.0, IBM, USA) will be used.

Key words: Stroke, mirror therapy, upper extremity, kinematic analysis

ELIGIBILITY:
Inclusion Criteria:1) to have a diagnosis of unilateral, ischemic or hemorrhagic, stroke for at least 6 months and at most 5 years ; 2) age between 30 and 80 years; 3) cognitive ability to follow the instructions of the study (Mini-Mental score ≥ 18 for schooling and ≥ 13 for illiterate);4) mild or moderate motor sensory impairment (Fugl-Meyer Assessment Scale - mild: 58-64 points, moderate: 39-57 points); 5) spasticity ≤ 2 in the flexor elbow and wrist muscles, and horizontal shoulder adductor (Modified Ashworth Scale); 6) muscle strength ≥ 3 in the flexor muscles of the shoulder, elbow and wrist, and elbow and wrist extensors (Kendall assessement).

-

Exclusion Criteria:

* Patients with visual impairment; history of severe depression or severe psychiatric disorder; other neurological or musculoskeletal disorders in the UE; visuospatial heminegligence; or pain file ≥ 4 on the compromised UE (Visual Analog Pain Scale), were excluded from the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-27 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Change Movement Cycle Time (MCT) | changes from baseline at 30 minutes after each session
  The time to perform the cycle of movement in seconds, which includes the going and return phase of the arm to the table
Change Index of Curvature (IC) | changes from baseline at 30 minutes after each session
  representative of the movement straightness during the going phase, an IC equal to 1 indicates a perfectly rectilinear motion
Change Average Jerk (AJ) | changes from baseline at 30 minutes after each session
  measure of the movement smoothness, this index decreases with increased smoothness
Change Mean Movement Velocity (MMV) | changes from baseline at 30 minutes after each session
  fingernail marker mean velocity during the going phase, an increased MMV indicates an improves task performance
Change Adjusting Sway (AS) | changes from baseline at 30 minutes after each session
  measure of the adjustments made to reach the target, decreases as the movement precision increases
Change Range of motion | changes from baseline at 30 minutes after each session
  Range of motion of shoulder (flexion/extension, abduction/adduction) and elbow (flexion/extension).

SECONDARY OUTCOMES:
Change Manual dexterity | changes from baseline at 30 minutes after each session
  Box and Block Test (BBT) was used to assess the gross manual dexterity. The test consists in moving, one by one, the largest possible number of blocks from one box compartment to the other, first with the uncommitted UE and then with the paretic UE. The recorded score is equivalent to the number of blocks moved from one side of the box to the other in 60 seconds
Change Spasticity of paretic upper extremity | changes from baseline at 30 minutes after each session
  The Modified Ashworth Scale (MAS) was used to assess spasticity, evaluating the resistance to passive movement. The patients stayed in a sitting position to the assessment of the muscle tone of the elbow flexors, wrist flexors and horizontal shoulder adductor of the paretic UE, with three mobilizations for each muscle group. Higher scores correspond to spasticity or increase in tone, while lower scores indicate normal muscle tone.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil